CLINICAL TRIAL: NCT00199771
Title: The Use of Hypertonic Saline Dextran in Cardiac Surgery Utilizing Cardio Pulmonary Bypass in Children Less Than 17 Weeks Old.
Brief Title: Hypertonic Saline Dextran in Pediatric Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: BioPhausia (Industry)
Responsible Party: Gunnar Bentsen / Consultant, Rikshospitalet-Radiumhospitalet HF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-HSD; S-01003 (ethics committee)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2008-01

CONDITIONS: Heart Defects, Congenital; Transposition of Great Vessels; Heart Septal Defects, Ventricular; Endocardial Cushion Defects
Keywords: Cardiac Surgery; Infant; Infant, Newborn; Hypertonic Solutions; Saline Solution, Hypertonic; Capillary leak; Inflammation Mediators
MeSH Terms: conditions — Heart Defects, Congenital; Transposition of Great Vessels; Heart Septal Defects, Ventricular; Endocardial Cushion Defects

INTERVENTIONS:
Drug: 7.5% NaCl in 6% dextran 70 solution

SUMMARY:
The purpose of this study is to determine whether infusion of hypertonic saline dextran attenuates the inflammatory response and the water overload, during and after major cardiac surgery in small children.

DETAILED DESCRIPTION:
After major cardiac surgery in small children, extravasation of fluid due to increased capillary leak has negative effect on haemodynamics and respiration. Inflammation cascades are activated by surgery and the use of cardio pulmonary bypass (CPB). We want to test whether a small infusion of 7.5% NaCl in 6% dextran solution before and after CPB reduces inflammatory activation by measuring the levels of interleukins 6 and 8 (IL-6, IL-8). We also measure extravascular lung water, fluid balance and weight during the first 24 hours post CPB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital heart defect undergoing surgery using cardio pulmonary bypass (CPB).
* Age below 17 weeks

Exclusion Criteria:

* Preoperative: organ failure (other than heart), serum sodium > 155 mmol/l, central venous pressure > 12 mmHg
* Perioperative: core temperature < 25 ºC on CPB, re-heparinization, re-operation

Max Age: 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14
Dates: Start 2003-06; Primary Completion 2004-12 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
IL-6 and IL-8 2 hours post CPB
Extra vascular lung water 2 and 24 hours post CPB

SECONDARY OUTCOMES:
Fluid balance
Weight gain
Cardiac output
Intrathorasic blood volume
Blood pressure during the first 24 hours post CPB

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Bentsen, MD, Principal Investigator — Oslo University Hospital